CLINICAL TRIAL: NCT00986570
Title: Phase III Open Label Clinical Trial to Assess Efficacy, Safety and Tolerability of Botulinum Toxin A (Xeomin®) in Treatment of Expression Wrinkles in the Upper Third of the Face
Brief Title: Clinical Trial to Assess Efficacy, Safety and Tolerability of Botulinum Toxin A (Xeomin®) in Treatment of Expression Wrinkles in the Upper Third of the Face
Acronym: XEO-001/07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEO-001/07
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Skin Aging
Keywords: Botulinum Toxin A; Wrinkles
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xeomin® (Experimental): Botulinum Toxin A
  Interventions: Biological: Botulinum Toxin A

INTERVENTIONS:
Biological: Botulinum Toxin A — 100 U DL50 lyophilized powder for reconstitution in 1 ml Saline Solution 0.9%.
  Other Names: Xeomin®

SUMMARY:
The purpose of this study is to determinate whether Xeomin® (Botulinum toxin Type A) is safe, effective and tolerable in woman aged 30 to 50 years old for treatment of mild, moderate or severe expression lines (wrinkles) in the upper third of the face. The main outcome was the change in appearance of the wrinkles two weeks (visit 3) after product application as compared with baseline assessment.

DETAILED DESCRIPTION:
Ageing is a dynamic and unchangeable process involving all individuals and affecting the several organic systems. This process is expressed through multiple symptoms and signs, the wrinkles and flaccidity being the most common and visible ones.

In both developed and emerging countries, the interest in skin ageing is, to a greater extent, the result of the progressive increase in the absolute number and the proportion of people experiencing the ageing process in the last century. The psychosocial, as well as the physiological effects of the skin ageing raised a huge demand for a better understanding of this process and, in particular, of the effective interventions.

The use of the botulinum toxin type-A (BTX/A) for aesthetic indication emerged as a result of the clinical observation of those patients treated for facial different dystonia and who presented additional improvement of their expression lines.

The expression lines are most easily noted on the upper third of the face, where surgical treatments are fully invasive and show lesser noticeable results. The upper third of the face was targeted for BTX/A treatment and reported in several scientific literature articles as well succeeded.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 to 50 years old, inclusive.
* Mild, moderate or severe expression wrinkles.
* Patients who had understood and signed the Informed Consent Form.

Exclusion Criteria:

* Subjects treated with botulinum toxin on the upper third of the face within the previous 6-month period;
* Former implantation of permanent material and surgery (scars).
* Use of any anticoagulant agent up to 7 days prior to the investigational product application;
* Concomitant use of aminoglycosides or of any other drug that may impair in the neuromuscular transmission;
* Coagulopathies and local inflammation/ infection at the application site.
* Diseases which do impact on the neuromuscular function, such as: myasthenia gravis, Eaton Lambert Syndrome;
* Pregnancy or breast feeding, women with potential to become pregnant or who do not agree to use an effective contraception method (Pearl Index < 1%);
* Allergy or known sensitivity to any of the components of the investigational drug;
* Subjects who were enrolled in other clinical trial for the last 12-month period prior to the present study, as per Resolution 251/97;
* Subjects who disagree with the study procedures, who do not sign the Informed Consent Form or who are not committed to participate in the trial.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Talarico, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo/Hospital São Paulo, São Paulo, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment : 01-Sep-2009 to 09-Feb-2010 Location: Outpatient clinic; Cosmiatry, surgery and oncology unit, Department of Dermatology, UNIFESP, Sao Paulo, Brazil
Groups:
- Xeomin®: Botulinum Toxin A in IM injections single dose as follows:
  24U in Orbicularis Oculorum (External area, 3 sites in each side) 20U in Glabella (5 sites) 8U in Frontal muscle (4 sites)
Period: Overall Study
Arm/Group | Xeomin®
Started | 121
Completed | 114
Not Completed | 7
Not completed — Lost to Follow-up | 6
Not completed — Potential bias for objective assessment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Xeomin®
Number analyzed (Participants) | 121
Age, Customized [Number; unit: participants]
  Between 30 and 50 years | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.52 (0.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121
  Male | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 121

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: Success has been defined as the reduction of any grade to a lower grade of expression wrinkles in the visit 3 (day 15) compared to the baseline assessment. The wrinkles will be classified according to the following: absence, mild, moderate, severe.
Time Frame: Baseline (pre-treatment) and Visit 3 (Day 15)
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Xeomin®
Number analyzed (Participants) | 121
% of participants | 89.08 [83.48 to 94.68]

ADVERSE EVENTS:
Arm/Group | Xeomin®
Serious Adverse Events (participants affected / at risk) | 1/121
Other Adverse Events (participants affected / at risk) | 94/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xeomin® (N=121)
Acute gastroenteritis (Gastrointestinal disorders) | 1 (1) — Required hospitalization. Not related to the study product.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xeomin® (N=121)
Eyelid edema (Skin and subcutaneous tissue disorders) | 2 (2) — Local adverse event
Injection-site bleeding (Surgical and medical procedures) | 39 (41)
Injection-site pain (Surgical and medical procedures) | 9 (9)
Injection-site pruritus (Surgical and medical procedures) | 4 (4) — Local adverse event
Deformity (Surgical and medical procedures) | 6 (6) — Local adverse event. Asymmetry after product injection.
Worsening of baseline wrinkles (Skin and subcutaneous tissue disorders) | 2 (2)
Site-injection edema (Surgical and medical procedures) | 1 (1)
Headache (Nervous system disorders) | 25 (25) — Three cases were not related and 22 cases were related to the study product.
Nausea (Gastrointestinal disorders) | 2 (2)
Sore throat (Infections and infestations) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No